CLINICAL TRIAL: NCT00547157
Title: A Phase 2 Randomized Trial of Radiotherapy Plus Panitumumab Compared to Chemoradiotherapy With Unresected, Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Radiotherapy Plus Panitumumab Compared to Chemoradiotherapy With Unresected, Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20062079; CONCERT2
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Cancer; Head and Neck Cancer; Oncology; Squamous Cell Carcinoma
Keywords: head and neck; squamous cell carcinoma; radiotherapy; chemoradiotherapy; panitumumab; locally advanced head & neck cancer; EGFr; epidermal growth factor receptor; SCCHN; locally advanced SCCHN; HNC; epidermal growth factor
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Panitumumab; Pharmaceutical Preparations; Cisplatin; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 1 CRT (Active Comparator): Cisplatin plus RT
  Interventions: Drug: Cisplatin
- ARM 2 PRT (Experimental): Panitumumab plus RT
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — Arm 2 consists of panitmumab plus RT
  Other Names: Panitumumab (drug)
  Arms: ARM 2 PRT
Drug: Cisplatin — Cisplatin
  Other Names: Cisplatin (Chemotherapy)
  Arms: ARM 1 CRT

SUMMARY:
The purpose of this study is to estimate, with pre-specified precision, the difference in local-regional control (LRC) rate at 2 years in subjects receiving chemoradiotherapy (CRT) or panitumumab plus radiotherapy (PRT) as first line treatment for locally advanced squamous cell carcinoma for the head and neck (SCCHN). A formal hypothesis will not be tested in this trial; however, the treatment arm difference in LRC rates at 2 years will be estimated.

DETAILED DESCRIPTION:
Primary Objective: To estimate, with pre-specified precision, the difference in local-regional control (LRC) rate at 2 years in subjects receiving chemoradiotherapy (CRT) or panitumumab plus radiotherapy (PRT) as first line treatment for locally advanced squamous cell carcinoma for the head and neck (SCCHN).

Secondary Objectives: To estimate the difference between 2 treatment regimens (CRT vs PRT) on other measures of clinical benefit, including LRC, overall response rate (ORR), progression-free survival (PFS), overall survival (OS); and safety.

Tertiary Objectives: To estimate the difference in health-related quality of life (HRQoL) and performance status in subjects receiving PRT or CRT.

Exploratory Objectives: To investigate potential biomarker development based on assessment of blood and tumor and the proposed mechanism of actions of study drugs. In addition, to investigate the effect of genetic variation in cancer genes and drug target genes on SCCHN and subject response to study drugs (separate informed consent required).

Hypothesis: A formal hypothesis will not be tested in this trial; however, the treatment arm difference in LRC rates at 2 years will be estimated.

Study Design: This is a phase 2, open-label, randomized, multicenter study. Eligible subjects will be randomized in a 2:3 ratio to either of the following regimens:

Arm 1 CRT:

* Accelerated fractionation RT: 70 to 72 Gy - delivered over 6 to 6.5 weeks
* Cisplatin: 100 mg/m2 (given on days 1 and 22 of RT) or

Arm 2 PRT:

* Accelerated fractionation RT: 70 to 72 Gy - delivered over 6 to 6.5 weeks
* Panitumumab: 9.0 mg/kg Q3W (given on days 1, 22, and 43 of RT)

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed SCC of the oral cavity, oropharynx, hypopharynx or larynx Stage III or Stage IVa-b (M0) disease according to the American Joint Committee on Cancer staging manual 6th edition (locally advanced) ECOG performance status of 0 or 1 Bidimensionally measurable disease >/= 10 mm in at least 1 dimension

Exclusion Criteria:

NO Primary tumor of the nasopharynx, sinuses, salivary gland, or skin NO Subjects requiring prophylactic tracheostomy NO Prior (or concomitant) malignancy (except non-melanomatous skin cancer or in situ cervical cancer), other than the study disease (SCCHN), unless treated with curative intent with no evidence of disease for >/= 3 years NO Prior treatment for locally advanced SSCHN NO Prior surgery for SCCHN (except nodal sampling or biopsy for study disease) NO Major surgery </= 28 days before randomization or minor surgery </= 14 days before randomization with the exception of feeding tube placement, dental extractions, central venous catheter placement, biopsies and nodal sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-11; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Giralt J, Trigo J, Nuyts S, Ozsahin M, Skladowski K, Hatoum G, Daisne JF, Yunes Ancona AC, Cmelak A, Mesia R, Zhang A, Oliner KS, VanderWalde A. Panitumumab plus radiotherapy versus chemoradiotherapy in patients with unresected, locally advanced squamous-cell carcinoma of the head and neck (CONCERT-2): a randomised, controlled, open-label phase 2 trial. Lancet Oncol. 2015 Feb;16(2):221-32. doi: 10.1016/S1470-2045(14)71200-8. Epub 2015 Jan 15. PMID 25596659
- [Background] Mesia R, Henke M, Fortin A, Minn H, Yunes Ancona AC, Cmelak A, Markowitz AB, Hotte SJ, Singh S, Chan AT, Merlano MC, Skladowski K, Zhang A, Oliner KS, VanderWalde A, Giralt J. Chemoradiotherapy with or without panitumumab in patients with unresected, locally advanced squamous-cell carcinoma of the head and neck (CONCERT-1): a randomised, controlled, open-label phase 2 trial. Lancet Oncol. 2015 Feb;16(2):208-20. doi: 10.1016/S1470-2045(14)71198-2. Epub 2015 Jan 15. PMID 25596660
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 152 subjects were enrolled with 90 subjects randomized to panitumumab plus radiotherapy arm, and 62 subjects randomized to chemoradiotherapy arm.
Groups:
- Panitumumab Plus Radiotherapy: Panitumumab (9.0 mg/kg day 1, day 22, day 43) plus Accelerated Fractionation Radiotherapy
- Chemoradiotherapy: Cisplatin (100 mg/m2 day 1 and day 22) plus Accelerated Fractionation Radiotherapy
Period: Overall Study
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Started | 90 | 62
Completed | 41 | 39
Not Completed | 49 | 23
Not completed — Other | 1 | 0
Not completed — Death | 38 | 18
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Administrative decision | 3 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Panitumumab Plus Radiotherpy: Consists of Panitumumab and Radiotherpy
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus Radiotherpy | Chemoradiotherapy | Total
Number analyzed (Participants) | 90 | 62 | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (8.3) | 57.4 (7.9) | 57.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 25
  Male | 72 | 55 | 127
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 00 | 0
  Black or African American | 0 | 0 | 0
  White | 88 | 60 | 148
  Hispanic or Latino | 2 | 2 | 4
Radiotherapy Delivery Modality [Number; unit: Participants]
  IMRT | 49 | 32 | 81
  3D-CRT | 41 | 29 | 70
  Missing | 0 | 1 | 1
Primary Tumor Site [Number; unit: Participants]
  Oropharynx/Larynx | 66 | 44 | 110
  Oral Cavity/Hypopharynx | 24 | 18 | 42
Nodal Status [Number; unit: Participants] — N0: No regional lymph node involvement; N+: Regional lymph node involvement
  Participants
    N0 | 11 | 7 | 18
    N+ | 79 | 55 | 134
Tumor Stage [Number; unit: Participants] — Tumor stage is determined according to TNM staging system. The tumor, node, and metastasis (TNM) staging system integrates clinical information, including that derived from endoscopy and radiological evaluation. Together the TNM classifications determine the overall clinical stage (I, II, III or IV).
  Participants
    T1-3 | 58 | 39 | 97
    T4 | 32 | 23 | 55

OUTCOME MEASURES:

1. Primary Outcome: Local Regional Control Rate at 2 Years
Description: Kaplan-Meier estimate of Local regional control rate at 2 years. Local regional control rate will be measured according to the investigator's assessment of disease status based on all available data (ie, from clinical examination, radiologic assessments, pathology reports, and autopsy reports).
Time Frame: from study day 1 to 2 years
Population: Efficacy Analysis Set
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 90 | 61
Proportion of Participants | 0.51 [0.40 to 0.62] | 0.61 [0.47 to 0.72]
Statistical Analysis 1: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; Risk Difference (RD) = -0.09, 95% CI 2-sided [-0.26 to 0.07] — difference is PRT - CRT

2. Secondary Outcome: Duration of Local Regional Control
Description: Time from study day 1 to the date of first local-regional failure or to death due to any cause (whichever occurs first)
Time Frame: maximum follow up time 46.2 months
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 90 | 61
months | 25.1 [12.0 to 36.0] | NA [14.4 to NA] — median time to event was not reached.
Statistical Analysis 1: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.0601, Regression, Cox; Hazard Ratio (HR) = 1.613, 95% CI 2-sided [0.980 to 2.656] — Hazard ratio is presented as panitumumab plus radiotherapy:chemoradiotherapy

3. Secondary Outcome: Progression-free Survival
Description: Time from first dose date till disease progression or death
Time Frame: maximum follow up time 46.2 months
Population: Efficacy analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 90 | 61
months | 17.3 [12.0 to 27.0] | NA [17.5 to NA] — median time to event was not reached.
Statistical Analysis 1: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.0259, Regression, Cox; Hazard Ratio (HR) = 1.731, 95% CI 2-sided [1.068 to 2.806] — Hazard ratio is presented as panitumumab plus radiotherapy:chemoradiotherapy

4. Secondary Outcome: Overall Survival
Description: Time from first dose date to death
Time Frame: maximum follow up time 46.2 months
Population: Efficacy Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 90 | 61
months | 41.7 [27.2 to NA] — The value is not estimable. | NA [NA to NA] — median time to event was not reached.
Statistical Analysis 1: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.1039, Regression, Cox; Hazard Ratio (HR) = 1.593, 95% CI 2-sided [0.909 to 2.793] — Hazard ratio is presented as panitumumab plus radiotherapy:chemoradiotherapy

5. Secondary Outcome: ORR by 6 Months - Central
Description: ORR is Objective Response Rate. Tumor assessments are based on central review of scans uisng a modification of the WHO criteria. Complete or partial response is considered as objective response.
Time Frame: From randomization to 6 months
Population: Evaluable for Central Tumor Response Analysis Set: the subset of subjects in the Efficacy Analysis Set with at least one bi-dimensionally measurable leasion at baseline using a modification of the WHO criteria per blinded central review.
Measure: Number (95% Confidence Interval); unit: Proporation of Participants
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 90 | 60
Proporation of Participants | 0.722 [0.618 to 0.812] | 0.767 [0.640 to 0.866]
Statistical Analysis 1: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.5744, Regression, Logistic; Odds Ratio (OR) = 0.791, 95% CI 2-sided [0.342 to 1.785] — The odd ratio is defined as the odds of having an objective response in the panitumumab plus radiotherapy arm relative to the odds in the chemoradiotherapy arm
Statistical Analysis 2: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; Difference in objective response rate = -0.044, 95% CI 2-sided [-0.187 to 0.112] — Difference is objective response rate in the panitumumab plus radiotherapy arm minus the rate in the chemoradiotherapy arm

6. Secondary Outcome: CRR by 6 Months - Central
Description: CRR is Complete Response Rate. Tumor assessments are based on central review of scans uisng a modification of the WHO criteria. Complete Response (CR) is defined as disappearance of all index lesions.
Time Frame: From randomization till 6 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Panitumumab Plus Radiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 90 | 60
Proportion of Participants | 0.144 [0.079 to 0.234] | 0.117 [0.048 to 0.226]
Statistical Analysis 1: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.8070, Regression, Logistic; Odds Ratio (OR) = 1.278, 95% CI 2-sided [0.438 to 4.043] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Panitumumab Plus Radiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; Difference in complete response rate = 0.029, 95% CI 2-sided [-0.103 to 0.141] — [estimate comment as in outcome 5, analysis 2]

ADVERSE EVENTS:
Time Frame: The median reporting period was around 74 days in the Panitumumab Plus Radiotherapy arm, and around 74 days in the Chemoradiotherapy arm.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. One Subject who was randomized to Panitumumab+Radiotherapy but received Chemotherapy+Radiotherapy was summarized under Chemotherapy+Radiotherapy arm. So the number of participants under Chemotherapy+Radiotherapy arm is 62 (61+1).
Arm/Group | Panitumumab Plus Radiotherapy | Chemotherapy Plus Radiotherapy
Serious Adverse Events (participants affected / at risk) | 30/89 | 25/62
Other Adverse Events (participants affected / at risk) | 88/89 | 61/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Radiotherapy (N=89) | Chemotherapy Plus Radiotherapy (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Aphagia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 3
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Death (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 6 | 6
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Sudden death (General disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Candidiasis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Weight decreased (Investigations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus Radiotherapy (N=89) | Chemotherapy Plus Radiotherapy (N=62)
Anaemia (Blood and lymphatic system disorders) | 6 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5
Ear pain (Ear and labyrinth disorders) | 6 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 6
Conjunctivitis (Eye disorders) | 6 | 0
Constipation (Gastrointestinal disorders) | 28 | 15
Diarrhoea (Gastrointestinal disorders) | 8 | 7
Dry mouth (Gastrointestinal disorders) | 30 | 21
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Dysphagia (Gastrointestinal disorders) | 64 | 39
Nausea (Gastrointestinal disorders) | 19 | 27
Odynophagia (Gastrointestinal disorders) | 33 | 22
Oral pain (Gastrointestinal disorders) | 6 | 7
Stomatitis (Gastrointestinal disorders) | 24 | 12
Vomiting (Gastrointestinal disorders) | 14 | 18
Asthenia (General disorders) | 11 | 14
Fatigue (General disorders) | 16 | 9
Mucosal inflammation (General disorders) | 54 | 42
Pain (General disorders) | 9 | 10
Pyrexia (General disorders) | 10 | 9
Candidiasis (Infections and infestations) | 3 | 4
Laryngitis (Infections and infestations) | 5 | 2
Oral candidiasis (Infections and infestations) | 12 | 11
Pharyngitis (Infections and infestations) | 8 | 2
Radiation mucositis (Injury, poisoning and procedural complications) | 7 | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 47 | 35
Weight decreased (Investigations) | 24 | 17
Decreased appetite (Metabolism and nutrition disorders) | 13 | 14
Dehydration (Metabolism and nutrition disorders) | 4 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Ageusia (Nervous system disorders) | 11 | 6
Dysgeusia (Nervous system disorders) | 18 | 21
Anxiety (Psychiatric disorders) | 5 | 5
Insomnia (Psychiatric disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Acne (Skin and subcutaneous tissue disorders) | 12 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 22 | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 15 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 0
Erythema (Skin and subcutaneous tissue disorders) | 13 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 0
Rash (Skin and subcutaneous tissue disorders) | 48 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.